CLINICAL TRIAL: NCT01717261
Title: Single Pre-Operative Radiation Therapy (SPORT) for Low Risk Breast Cancer
Acronym: SPORT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Michael Yassa, Radiation Oncologist, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12030
Record Dates: First submitted 2012-10-22; First posted 2012-10-30 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; early breast cancer; partial breast irradiation; preoperative radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Pre-Operative Radiation Therapy (Experimental)
  Interventions: Radiation: Single Pre-Operative Radiation Therapy

INTERVENTIONS:
Radiation: Single Pre-Operative Radiation Therapy — Dose escalation: 3 patients will receive 15 Gy in a single fraction. The following 3 patients will receive 18 Gy. The final 4 patients will receive 20 Gy.

SUMMARY:
The purpose of this study is to determine if partial breast irradiation administered in a single preoperative fraction is tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 60 years or older.
* Invasive ductal carcinoma.
* Unifocal disease.
* Tumors less than 2cm.
* No clinical evidence of nodal disease.
* Estrogen receptor status (ER) positive.
* Her2 negative.

Exclusion Criteria:

* Age less than 60 years.
* BRCA 1 and/or BRCA 2 mutation.
* Tumour histology limited to lobular carcinoma only.
* Neoadjuvant hormonal manipulation or chemotherapy.
* More than one primary tumour in different quadrants of the same breast.
* Inability to view tumor on imaging.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2018-12 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | 6 months
  Assess acute toxicity and wound healing complications from the preoperative radiation treatment as per NCI CTCAE Common Toxicity Scale.

SECONDARY OUTCOMES:
Chronic toxicity | 2 years
  Assess late-onset toxicity associated with a single fraction radiation treatement as per RTOG/EORTC Late Radiation Toxicity Scale
Cosmetic outcome | 5 years
  Cosmesis will be evaluated as per the EORTC Breast Cancer Cosmetic Rating scale.

OTHER OUTCOMES:
Ipsilateral breast cancer recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yassa, MD, Study Chair — Maisonneuve-Rosemon Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada